CLINICAL TRIAL: NCT07188285
Title: Mass Spectrometry-based Immune Profiling in Peripheral Blood of Autoimmune Diseases
Brief Title: Mass Spectrometry-based Immune Profiling in Autoimmune Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Zhejiang PuLuoTing Health Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, He Jing, Professor, Peking University People's Hospital
Other Study IDs: Immune profiling in AIDs
Record Dates: First submitted 2025-04-14; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erthematosus; Sjogren's Syndrome; Inflammatory Myopathies; Systemic Sclerosis (SSc); Vasculitis; Rheumatoid Arthritis (RA); Ankylosing Spondylitis; Osteoarthritis; Gouty Arthritis (GA); Psoriatic Arthritis (PsA); Healthy Controls
Keywords: autoimmune diseases; mass spectrometry
MeSH Terms: conditions — Myositis; Scleroderma, Systemic; Vasculitis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Osteoarthritis; Arthritis, Gouty; Arthritis, Psoriatic; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA anticoagulation and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The patients with active autoimmune diseases: The study will include patients with systemic lupus erythematosus, Sjogren's syndrome, inflammatory myopathy, systemic sclerosis, vasculitis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, osteoarthritis and gouty arthritis and healthy controls. About 50 patients of each type are required. The patients are in a state of disease activity and do not use biological agents.

SUMMARY:
Based on mass spectrometry flow method, this study analyzed the typing of new T, B, NK and DC cell subsets in peripheral blood of common autoimmune diseases and their correlation with disease activity, aiming at establishing an early screening and diagnosis model of autoimmune diseases.

DETAILED DESCRIPTION:
The study will include patients with systemic lupus erythematosus, Sjogren's syndrome, inflammatory myopathy, systemic sclerosis, vasculitis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, osteoarthritis and gouty arthritis and healthy controls. About 50 patients of each type are required. The patients are in a state of disease activity and do not use biological agents. Their peripheral blood will be detected by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, and aged 18-70 at the time of screening interview (inclusive).
2. The diagnosis of each disease meets the following standards - Systemic lupus erythematosus: 1997 ACR lupus classification standard

   * Behcet's disease: 2014 ICBD Behcet's disease classification standard
   * ANCA-associated vasculitis: 1990 American College of Rheumatology Classification Standard
   * Rheumatoid arthritis: 1987 ARA classification standard
   * Ankylosing spondylitis: new york standard revised in 1984
   * Sjogren's syndrome: 2016 ACR/EULAR Sjogren's syndrome classification standard
   * Inflammatory myopathy: Bohan recommended criteria in 1977
   * Systemic sclerosis: SSc standard formulated by American Rheumatology Association in 1980.
   * Psoriatic arthritis: CASPAR standard in 2006
   * Gouty arthritis: 1997 ACR gout classification standard
3. Disease activity status, each disease should meet the disease activity index;
4. Glucocorticoid (≤1mg/kg/d prednisone or other hormones with equivalent dose) was used before joining the group, and DMARDs (such as methotrexate, hydroxychloroquine, azathioprine, mycophenolate mofetil, leflunomide, cyclosporine, etc.) were allowed;
5. When participating in the trial, the patient must be informed in writing and hope that the patient can abide by the requirements of the research follow-up plan and other protocols.

   Exclusion Criteria:

1. Use IVIg or cyclophosphamide within 1.2 months, use other biological agents (infliximab, adalimumab, etanercept, anakinra, etc.) within 3 months, and use rituximab within 6 months; 2.1 months after receiving high-dose glucocorticoid (> 1 mg/kg/d). 3. Serious complications: including heart failure (≥ NYHA III), renal insufficiency (creatinine clearance rate ≤30 ml/min) and hepatic insufficiency (serum ALT or AST is greater than three times the normal upper limit, or total bilirubin is greater than the normal upper limit).

4. Other serious, progressive or uncontrollable hematological, gastrointestinal, endocrine, lung, heart, nerve or brain diseases (including demyelinating diseases, such as multiple sclerosis).

5. Suffering from serious infection (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, EB virus, tuberculosis infection), or being hospitalized due to infection, or using intravenous antibiotics to treat infection 2 months before the first dose of treatment.

6. Chest imaging showed abnormalities of malignant tumor or current active infection (including tuberculosis) within 3 months before enrollment.

7. Infected with HIV(HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If the serum is positive, it is recommended to consult a doctor with expertise in treating HIV or hepatitis C virus infection.

8. Any known malignant tumor or history of malignant tumor in the past 5 years. 9. Received any vaccination within 3 months before joining the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients are in a state of disease activity and do not use biological agents.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-16 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
proportion of immune cell subsets in peripheral blood. | through study completion, an average of 1 year
  Immune cell subsets include T cell, B cell, NK cell, Treg cell, Tfh cell, CLA+Treg cell, Tfr cell, Th1 cell, Th2 cell, Th17 cell and some unnamed cell subsets.

IPD SHARING:
Plan to Share IPD: No